CLINICAL TRIAL: NCT01714128
Title: Positron Emission Tomography (PET) With 18F-Fluoroestradiol (FES) as a Predictor of Response in Patients With Breast Cancer Scheduled to be Treated With MK-2206 in Combination With Either an Aromatase Inhibitor or Fulvestrant on NCI Protocol 8762
Brief Title: FES-PET for Patients Treated on NCI Protocol 8762
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Funding no longer available
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Farrokh Dehdashti, Professor of Radiology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dehdashti FES NCI#9167
Record Dates: First submitted 2012-10-17; First posted 2012-10-25 (Estimated); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
Keywords: NCI protocol #8762; Estrogen receptor positive breast cancer; recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — X-Rays; proto-oncogene protein c-fes-fps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Optional Diagnostic Imaging (Other): Optional diagnostic imaging FES-PET/CT imaging
  Interventions: Drug: Diagnostic Imaging ( 6α-[18F]fluoro-17β-estradiol (FES))

INTERVENTIONS:
Drug: Diagnostic Imaging ( 6α-[18F]fluoro-17β-estradiol (FES)) — FES-PET/CT imaging

SUMMARY:
A significant number of all invasive breast cancers are hormone sensitive and may be candidates for treatment with hormonal therapy.

This project will assess the ability and usefulness of imaging hormone-receptor status in breast cancer with positron emission tomography (PET) and 6α-[18F]fluoro-17β-estradiol (FES), an estrogen analogue in patients who are scheduled to be treated with hormonal therapy given in combination with a selective allosteric inhibitor of AKT protein kinase (MK2206) .

DETAILED DESCRIPTION:
Approximately 75% of all invasive breast cancers are hormone sensitive [estrogen-receptor positive (ER+) or progesterone-receptor positive (PR+)] and patients with such cancers are candidates for endocrine therapy. Endocrine therapy is a central component of the treatment of hormone-sensitive breast cancer in the adjuvant and, increasingly, neoadjuvant settings. Knowledge of hormone receptor expression is essential for selection of appropriate therapy. Measurement of hormone-receptor expression [estrogen receptor (ER) or progesterone receptor (PR)] using in vitro assays of the tumor tissue at the time of primary diagnosis is standard of clinical care. However, the presence of these hormone receptors predicts for clinical benefit in only 30-50% of women with advanced disease receiving first-line endocrine therapy and 15-30% receiving second-line therapy (1-3). Thus, the presence of a hormone receptor does not indicate that the receptor is functional and essential to the growth of the cancer cell, nor does it imply that interference with receptor function will result in tumor cell kill. There are several shortcomings of the in vitro assays and neither quantitative nor qualitative receptor assays performed on samples of tumor tissue completely predict the response to antiestrogen therapy in breast cancers. In addition, none of the current clinical tools (serologies, prognostic factors, or radiologic studies) can accurately predict for clinical benefit from endocrine therapy. Accordingly, better methods for predicting clinical response to antiestrogen therapy need to be developed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have agreed and signed consent to participate in NCI protocol 8762 and be scheduled to receive the first dose of MK-2206 in a minimum of 48 hours and a maximum of 30 days after the FES-PET/CT imaging.

   Note: Patients need to be on the endocrine agent for at least 1 week prior to the FES-PET/CT imaging.
2. Patients must have measurable disease (defined by RECIST criteria) or the presence of bone lesions if there is no measurable lesion.
3. Patient must be ≥ 18 years of age.
4. Patient must be able to tolerate and have no contraindication to FES-PET/CT imaging.
5. Patient must be able and willing to give informed consent.

Exclusion Criteria:

1. Patient must have no other active cancer at the time of study entry.
2. The research FES-PET/CT scan could not be scheduled more than 48 hours before starting therapy with MK-2206.
3. Patient cannot have received treatment for any other malignancy, with the exception of non-melanoma skin cancer, in the past 5 years.
4. Patients scheduled to receive chemotherapy as the primary source of treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
FES baseline tumor SUV measurement | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington Univesity in St. Louis
Locations (1):
- Mallinckrodt Institute of Radiology, St Louis, Missouri, United States